CLINICAL TRIAL: NCT03177239
Title: A Phase II Sequential Treatment Trial of Single Agent Nivolumab, Then Combination Ipilimumab + Nivolumab in Metastatic or Unresectable Non-Clear Cell Renal Cell Carcinoma (ANZUP1602).
Brief Title: Phase II Sequential Treatment Trial of Single Agent Nivolumab, Then Combination Ipilimumab + Nivolumab in Metastatic or Unresectable Non-Clear Cell Renal Cell Carcinoma (ANZUP1602)
Acronym: UNISoN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 1602
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Renal Cell Carcinoma; Papillary Renal Cell Carcinoma Type 1; Papillary Renal Cell Carcinoma Type 2; Chromophobe Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Xp11 Translocation Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Part 1: nivolumab 240mg IV q2w for a maximum of 12 months.
  Part 2; nivolumab 240mg IV q3w in addition to ipilimumab 1mg/kg q3w x 4 cycles Then nivolumab 240mg q2w for a maximum of 12 months.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Dosage Form: Nivolumab BMS-936558-01 Solution for Injection Potency: 100 mg (10 mg/mL) Primary Packaging: 10 mL vial Appearance: Clear to opalescent colourless to pale yellow liquid. May contain particles.
  Storage Condition: 2 to 8°C. Protect from light and freezing.
  Other Names: Opdivo
Drug: Ipilimumab — Dosage Form: Ipilimumab Solution for Injection Potency: 200 mg (5 mg/mL) Primary Packaging: 40 mL vial Appearance: Clear, colourless to pale yellow liquid. May contain particles. Storage Condition: 2 to 8°C. Protect from light and freezing.
  Other Names: Yervoy

SUMMARY:
This study aims to evaluate the safety, tolerability and effectiveness of new treatments for kidney cancer called Nivolumab and Ipilimumab. The study is in two parts; in the first instance patients receive nivolumab alone. If this treatment is not effective patients may move onto the second part of the trial, where they receive nivolumab + ipilimumab. There is no placebo.

The reason to offer one treatment alone, followed by two treatments together is that it is thought that the double treatment may have more side-effects, but also may be effective in people in whom the single first treatment (nivolumab alone) has not helped.

Nivolumab and ipilimumab are experimental treatments. This means that they are not an approved treatment for non-clear cell kidney cancer in Australia.

The purpose of this study is to test the effectiveness, safety, and tolerability of Nivolumab (also known as Opdivo or BMS-936558) and Ipilumumab (also known as MDX-010 or Yervoy). Nivolumab and ipilimumab are antibodies (a type of human protein) that are being tested to see if they will allow the body's immune system to work against tumour cells. The immune system is the body's defence against cancer, bacteria and viruses. The effectiveness of nivolumab and ipilimumab in cancer of the kidney will be assessed by measuring the size of patient tumours via CT scans.

Nivolumab and ipilimumab have been used alone or in combination in many other cancers, and are licenced for use in other cancers like advanced melanoma and bladder cancer in Australia. They have not been tested in people with non-clear cell kidney cancer.

About 85 participants with non-clear cell kidney cancer are expected to participate in this study, from Australia and New Zealand.

This research study has been initiated by Dr. Craig Gedye, is being conducted in collaboration with the Centre for Biostatistics and Clinical Trials (BaCT) and sponsored in Australia by the Australian and New Zealand Urogenital and Prostate (ANZUP) Cancer Trials Group Pty Ltd. Bristol Myers Squibb (BMS) is supplying the study drugs and grant funding for this research.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable, locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic nccRCC (both treatment-naïve or those treated with a VEGFR TKI or another systemic medical therapy). Non-clear cell histology including:

   * Papillary renal cell carcinoma (type 1)
   * Papillary renal cell carcinoma (type 2)
   * Other: including chromophobe renal cell carcinoma, pure sarcomatoid renal cell carcinoma, Xp11 translocation (TFE3+ IHC) carcinoma, other renal carcinoma NOS
2. Be ≥18 years of age on the day of signing informed consent
3. At least 1 target lesion according to RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. Adequate bone marrow function (should be performed within 14 days prior to registration and with values within the ranges specified below):

   * Haemoglobin ≥ 90g/L
   * Platelets ≥ 100x109/L
   * Neutrophil count ≥ 1.5x109/L
6. Adequate liver function (should be performed within 14 days prior to registration and with values within the ranges specified below):

   * Bilirubin ≤ 1.5 x upper limit of normal (ULN) except for participants with known Gilbert's syndrome who can have total bilirubin < 3.0 mg/dL
   * AST or ALT ≤ 3.0 x ULN (or ≤ 5.0x ULN in the presence of liver metastases)
7. Adequate renal function (should be performed within 14 days prior to registration and with values within the ranges specified below):

   * Creatinine ≤ 1.5x ULN OR
   * Creatinine clearance (CrCl) ≥ 30mL/min (use Cockcroft-Gault Formula)
8. Female participants of childbearing potential should have a negative urine or serum pregnancy within 24 hours prior to registering the patient. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female participants of childbearing potential should be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through to 5 months after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through to 7 months after the last dose of study therapy.
11. Able to provide a formalin-fixed paraffin embedded (FFPE) tumour block, representative of the participant's primary or metastatic disease (preferred), which must be forwarded to the Centre for Biostatistics and Clinical Trials (BaCT) within 10 working days post registration
12. Willing and able to start treatment within 14 days of registration, and to comply with all study requirements, including the timing and/or nature of the required treatment and assessments
13. Has provided signed, written informed consent.

Exclusion Criteria:

1. Urothelial or transitional cell carcinoma of the renal pelvis or ureter
2. Predominant clear cell renal cell carcinoma. A minority of clear cell histology (<50%) is acceptable, but there must be >50% non-clear cell histology predominant.
3. Participation in a study of an investigational agent within 30 days of registration.
4. Prior treatment with nivolumab, ipilimumab, or with any other anti-PD-1, anti-PD-L1, Anti-PD-L2, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways (NB Participant is eligible for Part 2 of the study if they took nivolumab monotherapy in Part 1 of the study).
5. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Any condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone or equivalent dose of alternative corticosteroid) or other immunosuppressive medications within 14 days of registration. Intranasal, inhaled or topical steroids are permitted in the absence of active autoimmune disease. Participants are permitted to enrol if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
7. Untreated brain or leptomeningeal metastases or current clinical or radiological progression of known brain metastases or requirement for steroid therapy for brain metastases. Participants with treated brain metastases are eligible if they have been stable and off steroids for ≥ 3 weeks.
8. Prior allogeneic organ transplant, inflammatory bowel disease, pneumonitis, tuberculosis, or primary immunodeficiency
9. Active infection requiring systemic therapy within 14 days before registration.
10. Receipt of live attenuated vaccination within 30 days of registration.
11. Life expectancy of less than 3 months.
12. Prior systemic therapy, surgery or radiation therapy within 4 weeks before registration.

    Note: If the participant has undergone major surgery, they must have recovered adequately before registration. Prior treatments with radiation therapy in the adjuvant and/or metastatic setting is permitted provided that therapy and is completed at least 14 days prior to the first dose of study drug and all treatment related adverse events are < Grade 1 at the time of registration.
13. History of another active malignancy within the previous 5 years, except for locally curable cancers that have been apparently cured, such as low-grade thyroid carcinoma, prostate cancer not requiring treatment (Gleason grade ≤ 6), basal or squamous cell skin cancer, superficial bladder cancer, melanoma in situ or carcinoma in situ of the prostate, cervix, or breast. Participants who have been free of other malignancies for ≥ 5 years prior to registration are eligible for this study.
14. Positive test for hepatitis B virus surface antigen (HBVsAg) or antibodies to hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
15. A history of other significant infection, including HIV. HIV testing is not mandatory unless clinically indicated.
16. Participants should be excluded if they have a history of allergy to study drug components, or a history of severe hypersensitivity reaction to any monoclonal antibody.
17. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol
18. Female patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The objective tumour response rate, as assessed by RECIST1.1 | Through study completion, on average 5 years.
  This is defined as the proportion of participants in the analysis set with a confirmed complete response (CR) or partial response (PR) divided by the number of participants in the analysis set.

SECONDARY OUTCOMES:
Duration of objective tumour response, as assessed by RECIST1.1 | Through study completion, on average 5 years.
  Measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that progressive disease is objectively documented.
Progression-free survival (PFS), as assessed by RECIST1.1 | Through study completion, on average 5 years.
  For Part 1, PFS is defined as the interval from date of registration to the date of first evidence of disease progression or death, whichever occurs first. For Part 2, PFS is defined as the interval from date of progressive disease on nivolumab monotherapy until the date of first evidence of disease progression or death, whichever occurs first.
Immune-related tumour response rate, as assessed by irRECIST. | Through study completion, on average 5 years.
  Defined as the proportion of participants in the analysis set with an immune related complete response (irCR), or immune related partial response (irPR), divided by the number of participants in the analysis set.
Immune-related disease control rate (irDCR6), as assessed by irRECIST. | At 6 months during treatment.
  For Part 1, irDCR6 is defined as an assessment of CR or iPR or iSD according to modified irRECIST. For Part 2, irDCR6 is defined in the same way except that the extent of disease defining the baseline tumour burden is measured at the date of disease progression on nivolumab monotherapy.
The number of patients alive at the end of the study, as assessed by date of death. | Through study completion, on average 5 years.
  Overall survival (OS) is defined as the time between the date of registration to part 1 of the study and the date of death due to any cause.
The number of patients with adverse events, particularly immune-related adverse events, that are related to study drug, as assessed and graded according to CTCAE v4.03. | From time of patient registration, until 30 days after the last dose of treatment.
The number of participants with permanent discontinuation of treatment or delays due to toxicity, as assessed and graded according to CTCAE v4.03. | From time of patient registration, until 30 days after the last dose of treatment.

OTHER OUTCOMES:
The biomarkers of response and resistance to anti-cancer treatments, as assessed by gene expression arrays, cytokine arrays, multiplex immunohistochemistry and mass cytometry on tissue and blood samples. | Through study completion, on average 5 years.

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (19):
  - Border Medical Oncology, Albury, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincents Hospital, Darlinghurst, New South Wales
  - Northern Cancer Institute, Frenchs Forest, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Tamworth Hospital - North West Cancer Centre, Tamworth, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Ashford Cancer Centre, Adelaide, South Australia
  - Ballarat Oncology & Haematology Services, Ballarat, Victoria
  - Box Hill Hospital - Eastern Health, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

REFERENCES:
- See also: Sponsor's website — http://www.anzup.org.au